CLINICAL TRIAL: NCT03864198
Title: Evaluation of Treatment With Trans-resveratrol, Folic Acid, Vitamin D, Vitamin B12 and B6 in Men With Infertility
Brief Title: To Evaluate the Effect of Reveratrol,Folic Acid, Vitamin D, Vitamin B12 and B6 in Male Infertility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Of Perugia (Other)
Collaborators: Ester Illiano, MD (Unknown)
Responsible Party: Principal Investigator, Elisabetta Costantini, Clinical Professor, University Of Perugia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESV1; 3310 (Registry Identifier: CEAS)
Record Dates: First submitted 2019-02-14; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Male Infertility
Keywords: Male infertility; Reveratrol; Vitamin B12; Vitamin B6; Folic acid
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genante (Tm) (Other): Genante tablets One tablet in the morning and one tablet in the evening for 3 months
  Interventions: Dietary Supplement: Genante

INTERVENTIONS:
Dietary Supplement: Genante — A dietary supplement for male infertility

SUMMARY:
The objective of this study is to evaluate the impact of the Genante(TM) on the spermiogram parameters in infertile male patients

DETAILED DESCRIPTION:
This is a single-centre prospective observational study. Twenty infertile male patients.

Inclusion criteria are:

Age:18-50 years oligozoospermia: < 5 million spermatozoa/mL; asthenozoospermia: < 32% progressive motile spermatozoa; teratozoospermia: < 4% normal forms.

Esclusion criteria:

Patients with azoospermia, who smoke, use drugs, drugs with proven fertility toxicity, exposed to any environmental or occupational toxic substances, radiation or heat; with orchitis secondary to mumps, sexually transmitted diseases, history of cryptorchidism, previous testicular torsion, genitourinary anomalies, alterations of the epididymis or deferens; and inguinal surgery

Pretreatment evaluation included:

Semen analysis Hormonal determinations:follicle-stimulating hormone (FSH) and luteinising hormone (LH) total Testosterone Total,estradiol, prolactina, 25-OH-Vitamin D3); scrotal ultrasound prostatic transrectal ultrasound

Outocmes measures (baseline, at 1 and 6 months):

* Semen volume (mL)
* Total sperm number (106/ejaculate)
* Sperm concentration (106/mL)
* Total motility (PR + NP)
* Progressive motility (PR, %)
* Vitality (live spermatozoa, %)
* Sperm morphology (normal forms, %)
* Ph
* FSH
* LH
* Testosterone totale
* Estradiol
* Prolactiona
* 25-OH-Vitamin D3
* scrotal ultrasound
* prostatic transrectal ultrasound

ELIGIBILITY:
Inclusion Criteria:

* male 18-50 years
* oligozoospermia: < 5 million spermatozoa/mL;
* asthenozoospermia: < 32% progressive motile spermatozoa;
* teratozoospermia: < 4% normal forms.

Exclusion Criteria:

* azoospermia
* smoke
* use drugs
* use drugs with proven fertility toxicity
* exposition to any environmental or occupational toxic substances
* exposition to radiation or heat
* orchitis secondary to mumps
* sexually transmitted diseases
* history of cryptorchidism
* previous testicular torsion
* genitourinary anomalies
* alterations of the epididymis or deferens
* inguinal surgery

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertile man
Enrollment: 20 (Estimated)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-03-20 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Semen volume at 1 month | 1 month
  semen volume in semen analysis
Change from 1month Semen volume at 6 months | 6 months
  semen volume in semen analysis
Change from baseline Total sperm number at 1 month | 1 month
  total sperm number in semen analysis
Change from 1 month Total sperm number at 6 months | 6 months
  total sperm number in semen analysis
Change from baseline Sperm concentration at 1 month | 1 month
  Sperm concentration in semen analysis
Change from 1 month Sperm concentration at 6 months | 6 months
  Sperm concentration in semen analysis
Change from baseline Total Motility at 1 month | 1 month
  total motility of spermatozoa in semen analysis
Change from 1 month Total Motility at 6 months | 6 months
  total motility of spermatozoa in semen analysis
Change from baseline Progressive motility at 1 month | 1 month
  Porgressive motility of spermatozoa in semen analysis
Change from 1 month Progressive motility at 6 months | 6 months
  Progressive motility of spermatozoa in semen analysis
Change from baseline Vitality at 1 month | 1 month
  live spermatozoa
Change from 1 month Vitality at 6 months | 6 months
  live spermatozoa
Change from baseline Sperm morphology at 1 month | 1 month
  normal forms of spermatozoa
Change from 1 month Sperm morphology at 6 months | 6 months
  normal forms of spermatozoa
Change from baseline FSH at 1 month | 1 month
  plasmatic evaluation of FSH
Change from 1 month FSH at 6 months | 6 months
  plasmatic evaluation of FSH
Change from baseline LH at 1 month | 1 month
  Plasmatic evaluation of LH
Change from 1 month LH at 6 months | 6 months
  Plasmatic evaluation of LH
Change from baseline Total testosterone at 1 month | 1 month
  plasmatic evaluation of total testosterone
Change from 1 month Total testosterone at 6 months | 6 months
  plasmatic evaluation of total testosterone
Change from baseline Prolactina at 1 month | 1 month
  plasmatic evaluation of prolactina
Change from 1 month Prolactina at 6 months | 6 months
  plasmatic evaluation of prolactina
Change from baseline 25-OH-Vitamin D3 at 1 month | 1 month
  plasmatic evaluation of 25-OH-Vitamin D3
Change from 1 month 25-OH-Vitamin D3 at 6 months | 6 months
  plasmatic evaluation of 25-OH-Vitamin D3
Change from baseline Scrotal ultrasound at 1 month | 1 month
  testis volume and vas deferens by ultrasound
Change from 1 month Scrotal ultrasound at 6 months | 6 months
  testis volume and vas deferens by ultrasound
Change from baseline Trans rectal Prostatic ultrasound at 1 month | 1 month
  prostate volume and morphology by ultrasound
Change from 1 month Trans rectal Prostatic ultrasound at 6 months | 6 months
  prostate volume and morphology by ultrasound
Change from baseline estradiol at 1 month | 1 month
  plasmatic evaluation of esatrdiol
Change from 1 month estradiol at 6 months | 6 months
  plasmatic evaluation of esatrdiol

CONTACTS AND LOCATIONS:
Overall Officials: Ester Illiano, MD, Study Director — University Of Perugia
Locations (1):
- Elisabetta Costantini, Terni, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agarwal A, Nallella KP, Allamaneni SS, Said TM. Role of antioxidants in treatment of male infertility: an overview of the literature. Reprod Biomed Online. 2004 Jun;8(6):616-27. doi: 10.1016/s1472-6483(10)61641-0. PMID 15169573
- [Background] Griveau JF, Le Lannou D. Reactive oxygen species and human spermatozoa: physiology and pathology. Int J Androl. 1997 Apr;20(2):61-9. doi: 10.1046/j.1365-2605.1997.00044.x. PMID 9292315
- [Background] Aitken RJ. Free radicals, lipid peroxidation and sperm function. Reprod Fertil Dev. 1995;7(4):659-68. doi: 10.1071/rd9950659. PMID 8711202
- [Background] de Lamirande E, Leclerc P, Gagnon C. Capacitation as a regulatory event that primes spermatozoa for the acrosome reaction and fertilization. Mol Hum Reprod. 1997 Mar;3(3):175-94. doi: 10.1093/molehr/3.3.175. PMID 9237244
- [Background] Hughes CM, Lewis SE, McKelvey-Martin VJ, Thompson W. The effects of antioxidant supplementation during Percoll preparation on human sperm DNA integrity. Hum Reprod. 1998 May;13(5):1240-7. doi: 10.1093/humrep/13.5.1240. PMID 9647554
- [Background] Erben RG, Soegiarto DW, Weber K, Zeitz U, Lieberherr M, Gniadecki R, Moller G, Adamski J, Balling R. Deletion of deoxyribonucleic acid binding domain of the vitamin D receptor abrogates genomic and nongenomic functions of vitamin D. Mol Endocrinol. 2002 Jul;16(7):1524-37. doi: 10.1210/mend.16.7.0866. PMID 12089348
- [Background] Hammoud AO, Meikle AW, Peterson CM, Stanford J, Gibson M, Carrell DT. Association of 25-hydroxy-vitamin D levels with semen and hormonal parameters. Asian J Androl. 2012 Nov;14(6):855-9. doi: 10.1038/aja.2012.77. Epub 2012 Oct 8. PMID 23042450
- [Background] Wong WY, Merkus HM, Thomas CM, Menkveld R, Zielhuis GA, Steegers-Theunissen RP. Effects of folic acid and zinc sulfate on male factor subfertility: a double-blind, randomized, placebo-controlled trial. Fertil Steril. 2002 Mar;77(3):491-8. doi: 10.1016/s0015-0282(01)03229-0. PMID 11872201
- [Background] Chen Q, Ng V, Mei J, Chia SE. [Comparison of seminal vitamin B12, folate, reactive oxygen species and various sperm parameters between fertile and infertile males]. Wei Sheng Yan Jiu. 2001 Mar;30(2):80-2. Chinese. PMID 11321956
- [Background] Das S, Lin HS, Ho PC, Ng KY. The impact of aqueous solubility and dose on the pharmacokinetic profiles of resveratrol. Pharm Res. 2008 Nov;25(11):2593-600. doi: 10.1007/s11095-008-9677-1. Epub 2008 Jul 16. PMID 18629618
- [Background] Amri A, Chaumeil JC, Sfar S, Charrueau C. Administration of resveratrol: What formulation solutions to bioavailability limitations? J Control Release. 2012 Mar 10;158(2):182-93. doi: 10.1016/j.jconrel.2011.09.083. Epub 2011 Sep 25. PMID 21978644
- [Background] Orihuela-Campos RC, Tamaki N, Mukai R, Fukui M, Miki K, Terao J, Ito HO. Biological impacts of resveratrol, quercetin, and N-acetylcysteine on oxidative stress in human gingival fibroblasts. J Clin Biochem Nutr. 2015 May;56(3):220-7. doi: 10.3164/jcbn.14-129. Epub 2015 Mar 28. PMID 26060353
- [Background] Liu J, Yi L, Xiang Z, Zhong J, Zhang H, Sun T. Resveratrol attenuates spinal cord injury-induced inflammatory damage in rat lungs. Int J Clin Exp Pathol. 2015 Feb 1;8(2):1237-46. eCollection 2015. PMID 25973008
- [Derived] Illiano E, Trama F, Zucchi A, Iannitti RG, Fioretti B, Costantini E. Resveratrol-Based Multivitamin Supplement Increases Sperm Concentration and Motility in Idiopathic Male Infertility: A Pilot Clinical Study. J Clin Med. 2020 Dec 11;9(12):4017. doi: 10.3390/jcm9124017. PMID 33322606